CLINICAL TRIAL: NCT05941988
Title: The Effect of Pre Grafting Partial Maxillary Expansion With Post Grafting Expansion Versus Pre Grafting Full Maxillary Expansion on the Stability and Bone Resorption in Secondary Unilateral Alveolar Cleft Grafting
Brief Title: Partial Maxillary Expansion With Post Grafting Expansion vs. Pre Full Maxillary Expansion in Secondary Alveolar Cleft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed fakhry, resident at oral and maxillofacial surgery department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 51853267
Record Dates: First submitted 2023-06-11; First posted 2023-07-12 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Alveolar Cleft

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre grafting partial maxillary expansion with post grafting expansion (Experimental): pregrafting partial maxillary expansion then grafting left bone to consolidate for 2 months followed by post grafting expansion till full arch alignment
  Interventions: Procedure: pre grafting partial maxillary expansion with post grafting expansion
- pre grafting full maxillary expansion (Active Comparator): pre grafting full maxillary expansion till full arch alignment then grafting and let bone to consolidate
  Interventions: Procedure: pre grafting partial maxillary expansion with post grafting expansion

INTERVENTIONS:
Procedure: pre grafting partial maxillary expansion with post grafting expansion — pre grafting partial maxillary expansion then anterior iliac grafting followed by 2 months period for consolidation then post grafting expansion till full arch alignment

SUMMARY:
Intermediate grafting with both pre- and post- grafting maxillary expansion with time span after grafting 6-8 weeks for consolidation and final retention for 3 months after finalization of expansion will get the advantages of both techniques combined.

DETAILED DESCRIPTION:
Secondary alveolar bone grafting (SABG) is an essential step in the overall management of Patients with cleft lip and palate (CLP). The numerous advantages of this procedure have been reported in the literature. However, resorption of the bone graft is a common situation, and the success of alveolar bone grafting (ABG) depends on several factors . The periodontal health of the surrounding graft tissues, the experience and ability of the surgeon and the timing of surgery are shown to be the most important factors determining success. Failure to rehabilitate the alveolar cleft may give rise to a variety of problems, including oronasal fistula, fluid reflux, speech pathology, impaired tooth eruption, lack of bone support for the anterior teeth, dental crowding, periodontal recession and eventual loss of teeth, and maxillary and facial asymmetry . Lack of alveolar bone also limits orthodontic treatment and/or prosthodontics rehabilitation. Post graft stimulation of maturation through remodeling of the graft is extremely important and is provided primarily by natural tooth eruption. Thus, the ideal time period for SABG is shown as to be the mixed dentition stage (9-12 years), just before the eruption of the permanent canine in line with the cleft. Timing of maxillary expansion in patients with cleft lip and palate is debated. Proponents of expanding the maxilla prior to secondary alveolar bone grafting state it is beneficial to align the segments prior to bone grafting better access for placement of the graft and working facility during surgery, However more recent literature shows maxillary expansion after secondary bone grafting is possible Advocates of expansion following grafting cite the advantages that bone consolidation is improved when the graft is placed under a dynamic load during healing and that there is a smaller soft tissue defect to close, less difficulty procuring an adequate volume of bone, and a narrower defect, which will regenerate bone more quickly and less possibility to induce oronasal fistula during maxillary expansion the study will change the concept of alveolar bone grafting in relation to maxillary expansion .just getting 5 mm minimal between two cleft edges and 2/3 of canine or lateral root has been formed and thin bone separate tooth from cleft defect the graft could be done

ELIGIBILITY:
Inclusion Criteria:

Patients with unilateral cleft alveolus with in the mixed dentition stage No intraoral soft and hard tissue pathology No systemic condition that contraindicate grafting

Exclusion Criteria:

* Local criteria:

  * poor oral hygiene
  * radiation therapy the head and neck cancers

Systemic criteria:

* immunity deficiency or hemorrhagic inherited diseases
* Bone pathology

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Bone volume change | 6 months
  bone volume is measured to ensure successful grafting

SECONDARY OUTCOMES:
presence of relapse of expansion | 8 months
  detection of any relapse after removal of maxillary expanders

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Uzel A, Benlidayi ME, Kurkcu M, Kesiktas E. The Effects of Maxillary Expansion on Late Alveolar Bone Grafting in Patients With Unilateral Cleft Lip and Palate. J Oral Maxillofac Surg. 2019 Mar;77(3):607-614. doi: 10.1016/j.joms.2018.07.022. Epub 2018 Jul 27. PMID 30138625
- [Background] Kaura AS, Srinivasa DR, Kasten SJ. Optimal Timing of Alveolar Cleft Bone Grafting for Maxillary Clefts in the Cleft Palate Population. J Craniofac Surg. 2018 Sep;29(6):1551-1557. doi: 10.1097/SCS.0000000000004680. PMID 29916970